CLINICAL TRIAL: NCT02873442
Title: Clinical Study Using Precision Cell Immunotherapy Combination With Transcatheter Arterial Chemoembolization in Advanced Liver Cancer
Brief Title: Precision Cell Immunotherapy Combined With TACE in Advanced Liver Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ningbo Cancer Hospital (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NBWYKY2016-06-005
Record Dates: First submitted 2016-08-15; First posted 2016-08-19 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-08

CONDITIONS: Precision Cell Immunotherapy; Transcatheter Arterial Chemoembolization; Advanced Liver Cancer
Keywords: Precision Cell Immunotherapy; Transcatheter Arterial Chemoembolization; Advanced Liver Cancer

ARMS (2):
- Precision cells combined with TACE (Experimental): Transcatheter Arterial Chemoembolization:
  patients will receive MMC,EADM hepatic arterial infusion,6 cycles. Precision Cells：After accepting concurrent TACE treatment,patients will receive 3 cycles of Precision Cells treatment
  Interventions: Procedure: TACE; Biological: Precision Cells
- Transcatheter Arterial Chemoembolization (Active Comparator): patients will receive MMC,EADM hepatic arterial infusion,6 cycles.
  Interventions: Procedure: TACE

INTERVENTIONS:
Procedure: TACE — Lipiodol 10-20ml,MMC 8～10mg,EADM20～ 40mg.According to tumor area of maximum diameter,0.1～0.2ml/cm2 Hepatic arterial infusion.
Biological: Precision Cells — DC cell suspension (1×107 DC+ physiological saline
  + 0.25% human bloodalbumin) 1ml for each infusion, subcutaneous injection for each infusion 3 cycles, each cycle received two infusions on day 19, 20; 40, 41; 61, 62. Precision Cell suspension (1-6×109 PMAT/PNAT + physiological saline + 0.25% human bloodalbumin) 300ml for each infusion, IV (in the vein) for each infusion 3 cycles, each cycle received one infusions on day 21, 42, 63.
  Arms: Precision cells combined with TACE

SUMMARY:
To evaluate the safety and effectiveness of cell therapy using precision cells Combined With TACE in Advanced Liver Cancer.

Eligibility:

Individuals greater than or equal to 18 years of age and less than or equal to 65 years of age who have been diagnosed with Advanced Liver Cancer.

DETAILED DESCRIPTION:
A total of 40 patients may be enrolled over a period of 1-2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18~65 years old, male or female;
2. Life expectancy≥6 months;
3. ECOG score: 0-3;
4. Advanced Malignancies (lung cancer, gastric cancer) were diagnosed by pathological or clinical physicians,and Diagnosis of hepatocellular carcinoma (HCC), surgery can not be performed but TACE treatment can be carried out;
5. Enough venous channel, no other contraindications to the separation and collection of white blood cells;
6. Laboratory examination: white blood cell≥3 x 10*9/L, blood platelet count≥60 x 10*/L, hemoglobin≥85g/L; lymphocyte count≥15%, total bilirubin≤100 mol/L; ALT and AST less than five times of the normal level; serum creatinine less than 1.5 times of the normal level；
7. Signed informed consent；
8. Women of child-bearing age must have evidence of negative pregnancy test and be willing to practice birth control after 2 weeks following the cells transfusion.

Exclusion Criteria:

1. Expected Overall survival < 3 months
2. The tumor size or quantity is not suitable for interventional treatment or portal vein tumor thrombus
3. Liver function is Childs Pugh C
4. Had received TACE therapy previously or in radiotherapy at present,or taking Sola Feeney
5. Other serious diseases:the heart,lung, kidney,digestive, nervous, mental disorders, immune regulatory diseases, metabolic diseases, infectious diseases, etc.
6. Unable or unwilling to provide informed consent, or fail to comply with the test requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-03 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2 years
Progress-free survival | 2 years

SECONDARY OUTCOMES:
Quality of life | 2 years
  Questionnaire will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Huajun Jin, Study Chair — Shanghai Cell Therapy Research Institute; Qijun Qian, Study Chair — Shanghai Cell Therapy Research Institute; Jiangtao Wang, Study Director — Ningbo No.5 Hospital (Ningbo Cancer Hospital)
Locations (1):
- Ningbo No.5 Hospital (Ningbo Cancer Hospital), Ningbo, Zhejiang, China